CLINICAL TRIAL: NCT00690495
Title: Prospective, Monocentric Controlled, Randomized, Double-blind Study to Compare the Two Different Propofol Emulsions Regarding Tolerability and Injection Pain During the Induction of Anesthesia in Adults
Brief Title: Use of a Modified Propofol Emulsion in Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: B. Braun Melsungen AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HC-G-H-0705
Record Dates: First submitted 2008-06-02; First posted 2008-06-04 (Estimated); Results first posted 2011-09-22 (Estimated); Last update posted 2012-01-05 (Estimated); Status verified 2012-01

CONDITIONS: Anesthesia
Keywords: Anesthesia; Induction; Pain
MeSH Terms: conditions — Pain | interventions — Propofol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Modified propofol (Propofol 0.5%)
  Interventions: Drug: Propofol
- 2 (Active Comparator): Propofol 1%
  Interventions: Drug: Propofol 1%

INTERVENTIONS:
Drug: Propofol — Propofol (drug), intravenous, induction of anesthesia
  Other Names: Modified propofol
  Arms: 1
Drug: Propofol 1% — Propofol (drug), intravenous, induction of anesthesia
  Other Names: Propofol-Lipuro 1%
  Arms: 2

SUMMARY:
The purpose of the study is to determine whether a modified propofol preparation shows any effect on the incidence of injection pain in adults undergoing elective surgery under general anesthesia.

Study hypothesis: The use of a modified propofol preparation will reduce the incidence of injection pain in the study group.

DETAILED DESCRIPTION:
Pain on injection is a most frequently reported side effect associated with the use of propofol for induction of anesthesia. Various measures have been taken to reduce the pain on injection, e.g. administration of lidocaine or fentanyl prior to propofol administration, mixture of lidocaine and propofol as well as cooling of the emulsion. Although pain on injection had been reduced with some of the above mentioned methods, they may not be regarded as a satisfactory solution of the problem.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adults, age ≥ 18 years and ≤ 80 years
* Anesthetic risk classified as ASA I-III
* Patients undergoing elective surgery under general anesthesia
* Signed informed consent

Exclusion Criteria:

* Simultaneous participation in another trial
* Known or suspected drug abuse
* Known hypersensitivity to Propofol, other ingredients of the emulsion, or to any other necessary co-medication
* Not allowed concomitant medication (psychopharmacologic agents, tranquilizers, or centrally active analgesics)
* Patients taking lipid lowering drugs
* History of decompensated renal failure
* History of severe hepatic dysfunction, hepatic cirrhosis
* Angiographically confirmed CHD (coronary heart disease) or cerebral ischemia
* History of convulsive disorders
* Decompensated cardiac insufficiency
* Hypovolemia
* Increased intracranial pressure
* Pregnancy (positive ß-HCG test) and lactation
* Emergency situation
* Patient who receives parenteral fat emulsion, e.g. intralipid
* Patients incapable of giving consent personally
* Venous access for induction of anesthesia not possible at dorsum of the hand or not dorsal

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2008-05; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Soltész, MD, PhD, Principal Investigator — Klinik für Anästhesie und operative Intensivmedizin, Klinikum Leverkusen gGmbH
Locations (1):
- Klinik für Anästhesie und operative Intensivmedizin, Klinikum Leverkusen gGmbH, Leverkusen, North Rhine-Westphalia, Germany

REFERENCES:
- [Derived] Soltesz S, Diekmann M, Mitrenga-Theusinger A, Keilen M, Molter GP. Reduced pain on injection with a 0.5% propofol emulsion during induction of anesthesia. Eur J Anaesthesiol. 2012 Mar;29(3):162-3. doi: 10.1097/EJA.0b013e32834cfa7d. No abstract available. PMID 22012178

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient in: 07.05.2008 Last patient out: 24.09.2008
Groups:
- Modified Propofol: Modified propofol (Propofol 0.5%)
- Propofol 1%: Propofol 1%
Period: Overall Study
Arm/Group | Modified Propofol | Propofol 1%
Started | 50 | 50
Primary Endpoint | 50 | 50
Completed | 50 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Modified Propofol | Propofol 1% | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 34 | 34 | 68
  >=65 years | 16 | 16 | 32
Age Continuous [Mean (Standard Deviation); unit: years] | 54.4 (14.6) | 55.2 (13.9) | 54.8 (14.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 15 | 26
  Male | 39 | 35 | 74
Region of Enrollment [Number; unit: participants]
  Germany | 50 | 50 | 100

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Expression of Pain During Injection
Time Frame: during first propofol bolus
Population: per protocol
Measure: Number; unit: participants
Arm/Group | Modified Propofol | Propofol 1%
Number analyzed (Participants) | 50 | 50
participants | 1 | 7

2. Secondary Outcome: Further Assessment of Injection Pain
Time Frame: during induction of anaesthesia and about 3 to 6 hours after end of anaesthesia
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Modified Propofol | Propofol 1%
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 44/50 | 26/50
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Modified Propofol (N=50) | Propofol 1% (N=50)
hypertriglyceridaemia (Metabolism and nutrition disorders) | 44 (44) | 26 (26)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less